CLINICAL TRIAL: NCT06188481
Title: Efficacy of Whole-body Electromyostimulation (WB-EMS) Training on Glycemic Control in People With Prediabetes: a Randomized Controlled Pilot-study
Brief Title: Efficacy of Whole-body Electromyostimulation (WB-EMS) Training in Participants With Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Mahdieh Shojaa, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WB-EMS
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group with WB-EMS Training (Other): The Intervention group receives 1.5 times a week WB-EMS training, wears an activity tracker for 16 weeks and completes 6 sessions of an evidence-based lifestyle education program.
  Interventions: Other: whole-body electromyostimulation training; Other: activity tracker; Other: evidence-based lifestyle education program
- Control group with activity tracker and evidence-based lifestyle education program (Other): The control group wears an activity tracker for 16 weeks and completes 6 sessions of an evidence-based lifestyle education program.
  Interventions: Other: activity tracker; Other: evidence-based lifestyle education program
- Control group with evidence-based lifestyle education program (Other): The control group completes 6 sessions of an evidence-based lifestyle education program.
  Interventions: Other: evidence-based lifestyle education program

INTERVENTIONS:
Other: whole-body electromyostimulation training — The duration of the intervention is 16 weeks, the training frequency is 1.5 times a week and the exercise program consists of 20 minutes.
  Arms: Intervention group with WB-EMS Training
Other: activity tracker — Participants wear the activity tracker on their wrist for the entire 16-week study period.
  Arms: Control group with activity tracker and evidence-based lifestyle education program; Intervention group with WB-EMS Training
Other: evidence-based lifestyle education program — Participants receive an evidence-based lifestyle education programme (6 x 20 minutes for the period of 3 month).

SUMMARY:
The goal of this pilot study is to assess the efficacy of the intervention (WB-EMS Training) in a sedentary group of adults with pre-diabetes and to estimate the potential effect sizes.

The main goals and questions it aims to answer are:

* Efficacy WB-EMS training in sedentary adults with pre-diabetes,
* Has WB-EMS training positive effects on HbA1c and other biomarkers?

Researchers will compare the intervention group with two control groups to see if WB-EMS training has effects on pre-diabetes.

DETAILED DESCRIPTION:
The study is planned as a randomized controlled pilot study. The intervention phase duration is set to 16 weeks. Prior to the study start, all subjects will be screened for their eligibility according to defined inclusion and exclusion criteria.

Sixty eligible sedentary individuals with pre-diabetes between the ages of 40 and 65 years will be randomised to one intervention group (n=20) and two control groups (n=20 each).

The main exercise intervention will be conducted via WB-EMS using a medical device approved system (miha bodytec®, Type II, Gersthofen, Germany). Participants in the intervention and one control group will receive an activity tracker (vivosmart 5, Garmin) to measure daily steps during the 16-week intervention phase. All study groups will further receive an evidence-based lifestyle education programme (6 x 20 minutes for 3 months), which provides education, information, and advice to prevent disease progression and improve quality of life and mobility.

During the baseline visit and after 16 weeks endpoint measurements incl. blood biomarkers, cardiometabolic and body composition parameters will be assessed. The intervention group will additionally attend a follow-up visit after 32 weeks and the parameters will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling sedentary (<20 min physical activity on <3 days/week) men and women aged 40-65 years without Diabetes Type 2
* elevated HbA1c levels (5.7%-6.4%),
* not functionally impaired (Short Physical Performance Battery (SPPB) ≥10)
* signed informed consent
* consent to use the WB-EMS and activity tracker

Exclusion Criteria:

* high-grade arrhythmia/VHF/SM carriers, heart failure >NYHA2, nephropathy (GFR<60),
* cognitive impairment
* Diabetes Type 2

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c in % | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Assessed via blood sample with finger stick technique

SECONDARY OUTCOMES:
Change from baseline in lipid profile in mg/dL | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Assessed via blood sample with finger stick technique. Includes LDL-cholesterol, HDL-cholesterol and triglycerides
Change from baseline in waist circumference in cm | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Assessed with a measure tape in the centre between the iliac crest and the lower edge of the last palpable rib
Change from baseline in body composition | Baseline, after 16 weeks of intervention and after follow-up 32 weeks (only intervention group)
  Lean body mass and total body fat in kg will be assessed with bioelectrical impedance analysis (BIA)
Change from baseline in depressive symptoms | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Standardized and validated questionnaire Patient Health Questionnaire consisting of 9 questions on depressive symptoms (PHQ-9) will be used. PHQ-9 is a self-reported questionnaire and is used to assess for the presence and severity of depressive symptoms. Possible score ranges from 0 (no depression) to 27 (severe depression).
Change from baseline in health-related quality of life | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Standardized and validated questionnaire WHO Health-Related Quality of Life (WHOQOL-BREF) consisting fo 26 questions on general quality of life will be used. The tool includes four domains: physical health, psychological health, social relationships, and environmental health; it also contains quality fo life and general health items. Each item of the WHOQOL-BREF is scored from 1 to 5 on a 5-point Likert scale. The scores are then transformed linearly to a 0-100-scale. A higher score indicates a higher quality of life.
Change from baseline in stress | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Standardized and validated questionnaire Perceived Stress Scale consisting of 10 questions about stress (PSS-10) will be used. In each questions, subjects are asked how often they felt a certain way on a 5-point scale from 1 for 'never' to 5 for 'very often'. The PSS score indicates levels of perceived stress, whereby higher scores indicate higher stress levels.
Change from baseline in well-being | Baseline, after 16 weeks of intervention and follow-up after 32 weeks (only intervention group)
  Standardized and validated questionnaire Secure Flourish Index (SFI) consisting of 12 questions on general well-being will be used. Each of the questions is assessed on a scale of 0 - 10. The SFI score is obtained by summing the scores from the 12 questions and results in a score from 0 - 120.

CONTACTS AND LOCATIONS:
Overall Officials: Mahdieh Shojaa, Dr., Principal Investigator — University Hospital Tuebingen/ Institute of Health Sciences/ Population-Based Medicine
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Said H. Screening for breast cancer. S Afr Med J. 1993 Oct;83(10):798. No abstract available. PMID 8093154
- [Background] Chakraborty R, Mukherjee B, Hati RN. Increase of the peroxidase activity of mouse submaxillary gland by reserpine. Life Sci. 1984 Nov 5;35(19):1913-9. doi: 10.1016/0024-3205(84)90471-5. PMID 6436608
- [Background] Martin HS, Kirk RM. Perforating bladder injury by impalement. Br J Clin Pract. 1966 Dec;20(12):652-3. No abstract available. PMID 5974506
- [Background] Bacon WL. Metabolism of lipid labeled very low density lipoprotein from laying turkey hens in laying turkey hens and immature turkeys. Poult Sci. 1981 Jul;60(7):1525-36. doi: 10.3382/ps.0601525. PMID 7322975
- [Background] Klasing KC, Jarrell VL. Regulation of protein degradation in chick muscle by several hormones and metabolites. Poult Sci. 1985 Apr;64(4):694-9. doi: 10.3382/ps.0640694. PMID 3889893
- [Background] Radouco-Thomas S, Grumbach P, Nosal G, Garcin F. [Toxicological study of some P factors]. Therapie. 1965 Jul-Aug;20(4):879-88. No abstract available. French. PMID 5845205
- [Background] Akine Y, Ogino T, Kajiura Y, Tsukiyama I, Egawa S, Yamada T, Tanemura K, Tsunematsu R, Ohmi K, Sonoda T, et al. Para-aortic nodal irradiation in the treatment of carcinoma of the uterine cervix: a report of 22 cases. Jpn J Clin Oncol. 1986 Dec;16(4):383-90. PMID 3795534
- [Background] van Buuren F, Horstkotte D, Mellwig KP, Frund A, Vlachojannis M, Bogunovic N, Dimitriadis Z, Vortherms J, Humphrey R, Niebauer J. Electrical Myostimulation (EMS) Improves Glucose Metabolism and Oxygen Uptake in Type 2 Diabetes Mellitus Patients--Results from the EMS Study. Diabetes Technol Ther. 2015 Jun;17(6):413-9. doi: 10.1089/dia.2014.0315. Epub 2015 Mar 3. PMID 25734937
- [Background] Miyamoto T, Fukuda K, Kimura T, Matsubara Y, Tsuda K, Moritani T. Effect of percutaneous electrical muscle stimulation on postprandial hyperglycemia in type 2 diabetes. Diabetes Res Clin Pract. 2012 Jun;96(3):306-12. doi: 10.1016/j.diabres.2012.01.006. Epub 2012 Jan 30. PMID 22296854
- [Background] Miyamoto T, Iwakura T, Matsuoka N, Iwamoto M, Takenaka M, Akamatsu Y, Moritani T. Impact of prolonged neuromuscular electrical stimulation on metabolic profile and cognition-related blood parameters in type 2 diabetes: A randomized controlled cross-over trial. Diabetes Res Clin Pract. 2018 Aug;142:37-45. doi: 10.1016/j.diabres.2018.05.032. Epub 2018 May 24. PMID 29802953
- [Background] Coughlin SS, Stewart J. Use of Consumer Wearable Devices to Promote Physical Activity: A Review of Health Intervention Studies. J Environ Health Sci. 2016 Nov;2(6):10.15436/2378-6841.16.1123. doi: 10.15436/2378-6841.16.1123. Epub 2016 Nov 30. PMID 28428979
- [Background] vanSonnenberg E, Wroblicka JT, D'Agostino HB, Mathieson JR, Casola G, O'Laoide R, Cooperberg PL. Symptomatic hepatic cysts: percutaneous drainage and sclerosis. Radiology. 1994 Feb;190(2):387-92. doi: 10.1148/radiology.190.2.8284385.
- [Background] Ellingson LD, Lansing JE, DeShaw KJ, Peyer KL, Bai Y, Perez M, Phillips LA, Welk GJ. Evaluating Motivational Interviewing and Habit Formation to Enhance the Effect of Activity Trackers on Healthy Adults' Activity Levels: Randomized Intervention. JMIR Mhealth Uhealth. 2019 Feb 14;7(2):e10988. doi: 10.2196/10988. PMID 30762582
- [Derived] Shojaa M, Knaub K, Schmitz N, Niess AM, Munz B, Rau S, Feit V, Mphepo W, Dingler R, Kemmler W. Effect of Whole-Body Electromyostimulation Training on Glycemic Control in People With Prediabetes: Protocol for a Pilot Randomized Controlled Trial Study. JMIR Res Protoc. 2025 Jun 24;14:e68761. doi: 10.2196/68761. PMID 40554784